CLINICAL TRIAL: NCT04723381
Title: A 15-Week Randomized Controlled Trial in Orthopedically Disabled Women
Brief Title: The Effect of Web Based Genital Hygiene Education Provided to Orthopedically Disabled Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siirt University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Sidar Gül, Principal Investigator, Siirt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1648
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Disability Physical; Genital Infection
Keywords: web based education; disabled women; genital hygiene; self care agency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Partivipants recieved web based genital hygiene education for seven week
  Interventions: Other: web based education
- Control (No Intervention): No intervention was applied to the women in the control group

INTERVENTIONS:
Other: web based education — Expert support and consultancy were received for the design and preparation of the web page.
  Arms: Experimental

SUMMARY:
The aim of this study is to determine the effect of web-based genital hygiene education provided to orthopedically disabled women on self care agency and genital hygiene behaviors.

DETAILED DESCRIPTION:
It was a randomized controlled trial. The women in the experimental group were given web-based genital hygiene education that continued for seven weeks. No intervention was applied to the women in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being orthopedically handicapped
* Being literate, being over the age of 18
* Having access to the internet
* Being able to use the internet/computer
* Being able to maintain genital hygiene individually.

Exclusion Criteria:

* The inability to use the internet
* Not being a member of the website
* Having mental retardation
* Being dependent on someone else to maintain genital hygiene (bedridden, with spasticity)
* No willing to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Introductory Questionnaire | Baseline
  The introductory questionnaire created for descriptive expressions
Change from the Baseline Self-Care Agency Scale Points at 7th and 15th weeks | Baseline, at the end of the 7th week, at the end of the 15th week
  Self-Care Agency Scale was used to determine the self-care skills and abilities of the participants. It is a 5-point Likert-type scale with 35 items. Each item of the scale is scored between 0 and 4 (0= very uncharacteristic of me, 4= very characteristic of me). In the scale, 8 items (3, 6, 9, 13, 19, 22, 26, and 31) are scored reversely (0= very characteristic of me, 4= very uncharacteristic of me). The scale is evaluated over 140 points. In evaluation, the score over 120 points is defined as high, the score between 82 and 120 points is defined as moderate, and the score below 82 points is defined as low.
Change from the Genital Hygiene Behavior Scale Points at 7th and 15th weeks | Baseline, at the end of the 7th week, at the end of the 15th week
  The Genital Hygiene Behavior Scale was used to determine the genital hygiene behaviors of the participants.It is a 5-point Likert-type scale with 23 items consisting of three sub-dimensions. The sub-dimensions of the scale are "General Hygiene (the first 12 items)", "Menstrual Hygiene (items between 13 and 20), and "Abnormal Finding Awareness (items between 21 and 23 )". Participants rate each item from 1 to 5 according to their suitability (1 = strongly disagree, 5 = Strongly agree). In the scale, 5 items (7, 14, 19, 20, 23) are scored reversely (1 = strongly agree, 5 = Strongly disagree). The highest score that can be obtained from the scale is 115 and the lowest score is 23. High scores indicate positive genital hygiene behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagul Yagmur, Prof, Study Director — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No